CLINICAL TRIAL: NCT00152074
Title: Effects of Modest Salt Reduction on Blood Pressure and Markers of Target Organ Damage in Patients With Untreated Essential Hypertension or Prehypertension
Brief Title: Salt Reduction on Blood Pressure and Cardiovascular Organ Damage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St George's, University of London (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CH/der/03.0214; N02034
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2006-09

CONDITIONS: Hypertension
Keywords: Blood pressure; Sodium; Dietary; Hypertension or prehypertension
MeSH Terms: conditions — Hypertension; Prehypertension

INTERVENTIONS:
Behavioral: Reduce salt intake

SUMMARY:
The purpose of this study is to determine the effect of a modest reduction in salt intake on blood pressure in white, black and Asian individuals with hypertension or prehypertension, and also to determine whether a modest reduction in salt intake has beneficial effects on the surrogate markers of target organ damage in cardiovascular disease.

DETAILED DESCRIPTION:
The average salt intake for adults in the UK is approximately 10-12 g/day. The current recommendations are to reduce salt intake to 5-6 g/day or less. Many randomised trials have shown that this reduction in salt intake has a significant effect on blood pressure, however, most previous trials were carried out in white individuals, fewer in blacks, and none in Asians.

Increasing evidence from epidemiological studies in humans and experimental studies in animals suggest that that our current high salt intake may have other harmful effects on cardiovascular health e.g. a direct effect on stroke, left ventricular hypertrophy, progression of renal disease and proteinuria independent of and additive to salt's effect on blood pressure. However, no well-controlled trials have studied whether a modest reduction in salt intake has beneficial effects on the surrogate markers of target organ damage in cardiovascular disease.

We propose to carry out a double-blind randomised trial to study the effects of a modest reduction in salt intake, as currently recommended, on blood pressure and target organ damage assessed by the measurements of 24 hour urinary albumin excretion, left ventricular mass, left ventricular diastolic function, pulse wave velocity and capillary density, in white, black and Asian individuals with hypertension or prehypertension.

Comparisons: Usual salt intake compared to reduced salt intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients with untreated essential hypertension or prehypertension (sitting systolic blood pressure between 120 and 170 mmHg and/or sitting diastolic blood pressure between 80 and 105 mmHg)
* Age 18 - 75 years.

Exclusion Criteria:

* Individuals younger than 18 or older than 75 years
* Individuals with severe hypertension i.e. blood pressure > 170/105 mmHg
* Individuals with any secondary cause of hypertension
* Individuals with impaired renal function with plasma creatinine greater than 150 umol/L
* Individuals with diabetes mellitus
* Individuals with malignancy or liver disease
* Individuals with ischaemic heart disease or heart failure
* Females who are pregnant or breast feeding or on the oral contraceptive pill.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2004-04; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure and markers of target organ damage at 6 weeks of usual salt intake vs those at 6 weeks of reduced salt intake.

SECONDARY OUTCOMES:
Comparisons among different ethnic groups in the changes in blood pressure and markers of target organ damage from week 6 of usual salt intake to week 6 of reduced salt intake.

CONTACTS AND LOCATIONS:
Overall Officials: Graham A MacGregor, MD, Principal Investigator — St George's, University of London
Locations (1):
- St. George's University of London,, London, United Kingdom

REFERENCES:
- [Derived] Chen L, He FJ, Dong Y, Huang Y, Wang C, Harshfield GA, Zhu H. Modest Sodium Reduction Increases Circulating Short-Chain Fatty Acids in Untreated Hypertensives: A Randomized, Double-Blind, Placebo-Controlled Trial. Hypertension. 2020 Jul;76(1):73-79. doi: 10.1161/HYPERTENSIONAHA.120.14800. Epub 2020 Jun 1. PMID 32475312
- [Derived] Chen L, He FJ, Dong Y, Huang Y, Harshfield GA, Zhu H. Sodium Reduction, Metabolomic Profiling, and Cardiovascular Disease Risk in Untreated Black Hypertensives. Hypertension. 2019 Jul;74(1):194-200. doi: 10.1161/HYPERTENSIONAHA.119.12880. Epub 2019 May 13. PMID 31079530